CLINICAL TRIAL: NCT05965531
Title: A Single-arm, Phase II Clinical Trial to Treat Locally Advanced, pMMR Rectal Cancer With Single-agent Trifluridine/Tipiracil Chemotherapy Plus Neoadjuvant Intensity-modulated Radiotherapy
Brief Title: Treating Locally Advanced Rectal Cancer With TAS-102 Chemotherapy Plus Neoadjuvant Radiotherapy
Acronym: TASLARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Chang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-087
Record Dates: First submitted 2023-07-14; First posted 2023-07-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; Trifluridine/Tipiracil; radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — trifluridine tipiracil drug combination; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: This phase 2 trial is an open-label, single-arm, non-comparative trial, in which all enrolled patients will receive neoadjuvant single-agent TAS-102 chemotherapy plus intensity-modulated radiotherapy, before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemo-radiotherapy with TAS-102 (Experimental): The patients in this group will all receive neoadjuvant treatment consisting of intensity-modulated radiotherapy and concurrent Trifluridine/Tipiracil (TAS-102). Then the ones evaluated to have a possibility of R0 resection will receive radical surgery, followed by 6 cycles of adjuvant XELOX (capecitabine plus oxaliplatin) chemotherapy.
  Interventions: Drug: Trifluridine/Tipiracil; Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — TAS-102 is given in a dose of 35 mg/m2, twice daily on the 1st to 5th and 8th to 12th days of the period of neoadjuvant radiotherapy.
  Other Names: TAS-102
Radiation: intensity-modulated radiotherapy — intensity-modulated radiotherapy

SUMMARY:
The goal of this Phase 2 trial is to evaluate a neoadjuvant treatment mode for locally advanced rectal cancer (LARC), consisting of radiotherapy and concurrent Trifluridine/Tipiracil (TAS-102). The main questions it aims to answer are: (i) whether TAS-102 is effective in treating LARC, when combined with radiotherapy; (ii) whether TAS-102 is safe in combination with radiotherapy. Participants will receive one cycle of TAS-102 chemotherapy and neoadjuvant radiotherapy based on intensity-modulated technique. Then the ones with a possibility of R0 resection will receive radical surgery followed by 6 cycles of adjuvant XELOX (capecitabine plus oxaliplatin) chemotherapy.

DETAILED DESCRIPTION:
The standard management recommended by the National Comprehensive Cancer Network for locally advanced rectal cancer (LARC) is neoadjuvant chemo-radiotherapy followed by surgery plus adjuvant chemotherapy or not. Currently, the regimens of neoadjuvant chemotherapy are based on fluorouracil or capecitabine. The therapeutic effects of these regimens are satisfactory, with a pathological complete response (pCR) and 3-year disease-free survival (DFS) rate of 14% and 68%. Addition of oxaliplatin has been proven to further improve the pCR and DFS rates, by the CAO/ARO/AIO-04, FOWARC and ADORE trials. However, the acute toxicities of fluorouracil and capecitabine remain as a concern. It was reported that the incidence of the grade 3/4 symptomatic toxicities brought by these two agents was nearly 15%. When combined with oxaliplatin, the incidence could rise to 25%. A special toxicity, hand-foot syndrome, was seen in 43-71% of the patients receiving capecitabine. It included blister, ulceration, numbness, pain and paresthesia, and seriously influenced the daily work and life of the patients. Trifluridine/Tipiracil (TAS-102) is a new generation of cytotoxic agent whose therapeutic effects in metastatic colorectal cancer have been confirmed by a series of large-scale, multicenter, randomized controlled trials. And the latest TASCO1 trial reported that TAS-102 exhibited a trend to improve overall survival, compared to capecitabine. Moreover, it could be well tolerated, with an incidence of grade 3/4 symptomatic toxicities of merely 1.5%. Until now, there was few study focusing on combination of TAS-102 and radiotherapy. This phase 2 trial intended to evaluate the therapeutic and adverse effects of TAS-102 concurrently with neoadjuvant radiotherapy, in a small patient cohort with LARC. The results might provide an effective and low-toxic choice which improves patients' experience of chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed rectal adenocarcinoma via biopsy
* Pretreatment clinical TNM stage as T3-4N0M0 or T1-4N1-2M0 (UICC TNM staging classification, version 8)
* Tumor with proficient DNA mismatch repair confirmed by immunohistochemical analysis
* Age between 18 and 75 years old
* Karnofsky performance score ≥ 70
* Distance from tumor lower margin to anal verge < 12 cm

Exclusion Criteria:

* Inguinal lymph node metastasis
* Multiple primary colorectal cancer
* Complete obstruction or perforation
* Uncontrolled tuberculosis, AIDS or mental diseases
* Severe cardiac, renal, hepatic or hematopoietic dysfunctions unsuitable for chemotherapy or radiotherapy
* Prior history of other malignancies with 5 years, except cured cervical carcinoma in situ and skin basal cell carcinoma
* Prior history of rectal surgery, pelvic radiotherapy or chemotherapy
* Pregnant or lactating women
* Other situations for which the investigators consider a patient inappropriate to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | One week after surgery
  The percentage of the patients complete R0 resection and attain a tumor regression grade of 1-4 (Mandard's 5-tier standard) in postsurgical pathologic examination

SECONDARY OUTCOMES:
Pathological complete response rate | One week after surgery
  The percentage of the patients complete R0 resection and attain a complete remission of both primary tumor and regional lymph nodes in postsurgical pathologic examination
The incidence of grade 3/4 toxicities | Once a week during the period of neoadjuvant treatment
  The percentage of the patients undergo any grade 3/4 toxicity during neoadjuvant treatment, based on the Common Terminology Criteria for Adverse Events
The incidence of grade 3/4 complications | The period from the date of radical surgery to the 90th day after surgery
  The percentage of the patients undergo any grade 3/4 surgery-related complication, based on the Clavien-Dindo classification.
Disease-free survival | When all the patients are followed-up for 1, 2 and 5 years
  The percentage of the patients survive without local recurrence or distant metastasis after a time period, from pathological diagnosis
Overall survival | When all the patients are followed-up for 1, 2 and 5 years
  The percentage of the patients survive after a time period, from pathological diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China